CLINICAL TRIAL: NCT05808751
Title: Clinical Cardiac Rehabilitation Registry Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-1785
Record Dates: First submitted 2023-03-01; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establish an electronic cardiac rehabilitation patient registration system and clinical database, carry out prospective cohort follow-up and observation of cardiovascular disease (CVD) patients receiving cardiac rehabilitation in inpatients and outpatients, collect risk factors, diagnosis and treatment status, rehabilitation diagnosis and treatment, clinical outcomes and follow-up results, and establish a short-term and long-term follow-up mechanism.

DETAILED DESCRIPTION:
Establish an electronic cardiac rehabilitation patient registration system and clinical database, carry out prospective cohort follow-up and observation of cardiovascular disease (CVD) patients receiving cardiac rehabilitation in inpatients and outpatients, collect risk factors, diagnosis and treatment status, rehabilitation diagnosis and treatment, clinical outcomes and follow-up results, and establish a short-term and long-term follow-up mechanism. Through the real world clinical practice data of cardiac rehabilitation of CVD patients, describe the population and disease characteristics of cardiac rehabilitation patients, the provision of cardiac rehabilitation services and the influencing factors; Analyze and study the key technologies of clinical cardiac rehabilitation, evaluate the implementation quality of cardiac rehabilitation, improve the clinical pathway of cardiac rehabilitation, and optimize the service process.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older.
2. Patients receiving inpatient cardiac rehabilitation, and/or participating in outpatient cardiac rehabilitation.
3. All cases selected were in New York Heart Association (NYHA) cardiac function class II and below.
4. Normal troponin.
5. Patients with some ability to communicate and understand.
6. have signed an informed consent form. -

Exclusion Criteria:

1. Subjects who are participating in clinical trials of other drugs or devices.
2. Patients with NYHA cardiac function class III or higher.
3. Mentally impaired, or unable to communicate effectively with investigators.
4. Refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CVD who received inpatient cardiac rehabilitation at Fu Wai Hospital and those who participated in outpatient cardiac rehabilitation at the Cardiac Rehabilitation Center of Fu Wai Hospital after discharge from the hospital
Sampling Method: Probability Sample
Enrollment: 2081 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause and attributed deaths | 1-year and 2-year
  All-cause and attributed deaths during hospitalization and follow-up of CVD patients
Major adverse cardiovascular events (MACE) occurrence | 1-year and 2-year
  Major adverse cardiovascular events (MACE) occurrence include cardiovascular death, non-fatal stroke, non-fatal myocardial infarction (MI), and ischemia-driven revascularization.

SECONDARY OUTCOMES:
Cardiopulmonary function and quality of life | 1-year and 2-year
  Cardiopulmonary function and quality of life in cardiac rehabilitation patients during the follow-up period
Participation and adherence | 1-year and 2-year
  Participation and adherence in outpatient cardiac rehabilitation.
Medical costs of cardiac rehabilitation patients during hospitalization and up to 2 years after discharge. | 1-year and 2-year
  Medical costs of cardiac rehabilitation patients during hospitalization and up to 2 years after discharge.
Proportion of different comorbidities, interactions and prognosis in CVD. | 1-year and 2-year
  Proportion of different comorbidities, interactions and prognosis in CVD.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Feng, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No